CLINICAL TRIAL: NCT02616289
Title: Topical Emollient Therapy in the Management of Severe Acute Malnutrition: A Randomized Controlled Clinical Trial in Bangladesh
Brief Title: Emollient Therapy for Severe Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: GlaxoSmithKline (Industry); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-15101
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Child Malnutrition; Malnutrition in Children; Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition | interventions — Emollients

STUDY DESIGN:
Intervention Model Description: Clinical Trial in two treatment arms
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Emollient (Experimental): Topical emollient (Sun Flower seed oil) in addition to routine standard of care for severe acute malnutrition.
  Interventions: Other: Topical emollient (Sun Flower seed oil)
- Control (No Intervention): Routine Standard of care only for severe acute malnutrition.

INTERVENTIONS:
Other: Topical emollient (Sun Flower seed oil) — 3 g of oil per kg of infant's weight at study entry of Sunflower Seed oil (SSO) will be applied three times per day at regularly spaced intervals (8-hour intervals) for 10 days. Oil will not be applied to the face (to avoid the possibility of any accidental aspiration or ingestion), ears or under the hairline. Care will be taken to not injure the skin during the massage treatment. The child's anal area will be washed prior to application to avoid the spread fecal flora from the anal region (to which the oil will be applied to last). Prior to bathing the child a minimum of 3-4 hours should have elapsed following the application of the SSO. The amount of oil required will be calculated based on the child's weight and the required amount weighed out each time.
  Arms: Emollient

SUMMARY:
The investigators hypothesize that the absorption of topically applied EFA-containing emollient (SSO) into the skin and thence into the bloodstream in children with SAM will improve skin barrier function and accelerate weight gain and clinical rehabilitation beyond that possible through normal standard-of-care

DETAILED DESCRIPTION:
A child with SAM, in addition to wasting will often present with infection, hypothermia, dehydration and electrolyte imbalance - complications attributable, at least in part, to compromised skin barrier function. Essential fatty acid (EFA)-containing emollients such as sunflower seed oil (SSO) have been shown to augment skin barrier function, reduce transepidermal water loss (TEWL) and risk of bloodstream infection and mortality, and promote weight gain in preterm infants. Recent research from rural Bangladesh showed very low levels of EFAs in young children in the general population. It is believed that EFA levels will be further depleted in children with SAM. So the investigators aim to demonstrate the feasibility of topical applications of SSO to children with SAM, and to measure clinical impact of emollient therapy with SSO on skin barrier function, skin condition, EFA levels in blood, weight gain, co-morbidities (e.g., pneumonia, sepsis), and time to complete acute rehabilitation from SAM, in addition to the benefits of normal standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian is willing and able to provide written informed consent for the subject to take part in the trial and comply with an inpatient stay of at least 10 days.
* Children aged 2-24 months inclusive diagnosed with SAM (weight-for-length Z score <-3 or bilateral pedal edema) admitted in the Dhaka Hospital of icddr,b, Dhaka, Bangladesh
* Willing to suspend usual home skin care treatments for the duration of study

Exclusion Criteria:

* Consent refusal
* Life threatening health conditions such as septic shock and altered consciousness on admission; congenital problems (congenital heart disease or known metabolic disorders, chromosomal abnormalities, renal failure, etc.); any known chronic disease including tuberculosis, HIV infection
* History of drug or other allergy or any condition that may complicate the interpretation of safety or efficacy such as dermatitis which, in the opinion of the investigator, contraindicates participation in the trial, or know hypersensitivity to SSO
* The child is in care (no longer looked after by their parent or legal guardian)
* Participation in another study

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
changes of body weight | Baseline and 10th day
  Body weight will be measured after 10 days of intervention

SECONDARY OUTCOMES:
Time to discharge from acute illnesses | through study completion, an average of 5 days
  Time to discharge from acute illnesses like, diarrhea, pneumonia, enteric fever etc which usually associated with severe acute malnutrition.
Reduction of rate of nosocomial infections between cases and controls | through study completion, an average of 10 days
  Reduction of rate of nosocomial infections between cases and controls
Reduction in TEWL | baseline and 10th day
  Reduction in trans-epidermal water loss (TEWL) which will be measured by Tewameter
Serum CRP level | Baseline and 10th day
  Serum CRP level will be assessed before and after the intervention to know the potential impact of the intervention on this change.
Serum Cytokines level | Baseline and 10th day
  Serum Cytokines (inflammatory) level will be assessed before and after the intervention to know the potential impact of the intervention on these changes.
Serum essential fatty acids (EFAs) level | Baseline and 10th day
  Serum EFAs level will be assessed before and after the intervention to know the potential impact of the intervention on these changes.
Skin condition changes | Baseline and 10th day
  Clinical improvement of skin conditions will be measured by a predefined skin scoring system where the value of the score increase proportionately (score '0' in normal skin condition) with the skin changes. Investigators will compare the score with baseline after intervention among the groups.

CONTACTS AND LOCATIONS:
Overall Officials: K M Shahunja, MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital, icddr,b, Dhaka, Bangladesh

REFERENCES:
- [Derived] Fischer N, Darmstadt GL, Shahunja KM, Crowther JM, Kendall L, Gibson RA, Ahmed T, Relman DA. Topical emollient therapy with sunflower seed oil alters the skin microbiota of young children with severe acute malnutrition in Bangladesh: A randomised, controlled study. J Glob Health. 2021 Jul 17;11:04047. doi: 10.7189/jogh.11.04047. eCollection 2021. PMID 34386216
- [Derived] Shahunja KM, Sevin DC, Kendall L, Ahmed T, Hossain MI, Mahfuz M, Zhu X, Singh K, Singh S, Crowther JM, Gibson RA, Darmstadt GL. Effect of topical applications of sunflower seed oil on systemic fatty acid levels in under-two children under rehabilitation for severe acute malnutrition in Bangladesh: a randomized controlled trial. Nutr J. 2021 Jun 6;20(1):51. doi: 10.1186/s12937-021-00707-3. PMID 34092255
- [Derived] Shahunja KM, Ahmed T, Hossain MI, Mahfuz M, Kendall L, Zhu X, Singh K, Crowther JM, Singh S, Gibson RA, Darmstadt GL. Topical emollient therapy in the management of severe acute malnutrition in children under two: A randomized controlled clinical trial in Bangladesh. J Glob Health. 2020 Jun;10(1):010414. doi: 10.7189/jogh.10.010414. PMID 32509290